CLINICAL TRIAL: NCT02927015
Title: Glucose Response From Antioxidant Rich Potato Chips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Richard Mattes, Prof. Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 055-043
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Glycemic Response

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Purple Majesty potato chips (Experimental): Purple Majesty potato chips
  Interventions: Other: Purple Majesty potato chips
- Mountain Rose potato chips (Experimental): Mountain Rose potato chips
  Interventions: Other: Mountain Rose potato chips
- White potato chips (Experimental): White potato chips
  Interventions: Other: White potato chips
- Crackers (Experimental): Crackers
  Interventions: Other: Crackers

INTERVENTIONS:
Other: Purple Majesty potato chips — Purple Majesty potato chips
  Arms: Purple Majesty potato chips
Other: Mountain Rose potato chips — Mountain Rose potato chips
  Arms: Mountain Rose potato chips
Other: White potato chips — White potato chips
  Arms: White potato chips
Other: Crackers — Crackers
  Arms: Crackers

SUMMARY:
Assess impact of potato phytochemical on post-prandial gastric emptying and glucose release from products in a pilot human study.

DETAILED DESCRIPTION:
Preclinical data obtained using an Caco-2 intestinal cell model and enzyme assays suggest phenolic-rich potato extracts decrease intestinal glucose transport. The aim is to determine if these effects extend to the the an in vivo situation. Specifically, the glycemic response following consumption of phenolic rich pigmented potatoes compared to white potatoes with lower phenolic content will be measured. Gastric emptying will also be measured to show the effects are in fact due to rate of carbohydrate digestion and intestinal glucose transport and not gastric emptying rate.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 non-smoker

Exclusion Criteria:

* BMI outside 18-25 smoker previous gastrointestinal disease or other disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | up to 2 hours
  blood taken at 10, 20, 30, 60, and 120 minutes by finger prick
Gastric emptying | up to 4 hours
  Breath Hydrogen concentrations will be measured every 15 minutes for 4 hours

IPD SHARING:
Plan to Share IPD: No